CLINICAL TRIAL: NCT05229133
Title: A Multicentre, Prospective, Single-arm Clinical Trial to Evaluate Efficacy and Safety of Femtosecond Laser Corneal Lenticule Extraction for Advanced Refractive Correction (CLEAR) in Myopia and Astigmatism in Chinese Population
Brief Title: Efficacy and Safety of CLEAR in Myopia and Astigmatism in Chinese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziemer Ophthalmic Systems AG (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPFLM-0008-CN-01
Record Dates: First submitted 2021-12-22; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-12

CONDITIONS: Myopic Astigmatism
Keywords: CLEAR; Ziemer; FEMTO LDV; Lenticule; Myopic astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refractive correction using CLEAR (Experimental): Subjects 18+ years old with myopic (-0.50 to -10.00 D) astigmatism (up to -5.00 D) treated bilaterally with FEMTO LDV Z8 using CLEAR application.
  Interventions: Device: CLEAR

INTERVENTIONS:
Device: CLEAR — FEMTO LDV Z8 Surgical Laser is intended for use in Corneal Lenticule Extraction for Advanced Refractive correction (CLEAR), also called Curved Lamellar Resection (CLR), for the reduction or elimination of myopia from -0.50 D to -10.00 D, with astigmatism of 0 D to -5.00 D or without astigmatism, and MRSE of -0.50 D to -12.50 D in the eye to be treated in patients who are 18 years of age or older with documentation of stable manifest refraction over the past year as demonstrated by a change in sphere and cylinder of ≤ 0.50 D in magnitude.
  Other Names: Corneal lenticule extraction for advanced refractive correction

SUMMARY:
In this multicenter, prospective, interventional, single-arm clinical trial, the aim is to determine safety and efficacy of CLEAR using the FEMTO LDV Z8 in Chinese patients in China.

The primary objective is to evaluate the visual outcome after CLEAR using the FEMTO LDV Z8 in myopia and astigmatic myopia at the time point, when stability of manifest refraction spherical equivalent (MRSE) is reached.

The corresponding hypothesis is that the percentage of treated eyes with satisfactory Uncorrected Distance Visual Acuity (UCDVA) at the point when stability of MRSE is reached after CLEAR is at least 85% of all treated eyes. This hypothesis has been chosen in line with the recommendations of the "Checklist of Information Usually Submitted in an Investigational Device Exemptions (IDE) Application for Refractive Surgery Lasers" issued by the FDA.

The secondary objectives are to evaluate the efficacy and safety with respect to stability, predictability, device defects and adverse events of CLEAR using the FEMTO LDV Z8 in myopia and astigmatic myopia during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Medically suitable for corneal refractive surgery
2. Signed informed consent form
3. Age ≥ 18 years
4. Pre-operative BCVA ≥ 5.0 (corresponding to 20/20 as per Snellen chart lines)
5. Myopia sphere from -0.5 D to -10.00 D
6. Maximum cylinder diopter of -5.00 D
7. Maximum resulting MRSE of -12.5 D
8. Calculated residual stromal thickness ≥ 250 microns
9. Non-contact IOP < 21mmHg
10. Stable refraction for the past year, as demonstrated by a change in manifest refraction spherical equivalent (MRSE) of ≤ 0.50 D
11. A difference between cycloplegic refraction spherical equivalent and MRSE < 0.75 D.
12. For contact lens wearers (where applicable) after pre-operative stop of contact lens wear: Stable refraction (within ±0.5 D), as determined by MRSE, on two consecutive examinations at least 1 week apart.
13. Patient willing and able to return to the study site for the follow-up visits, in the judgement of the investigator.

Exclusion Criteria:

1. Wearing of contact lenses pre-operatively i) soft contact lenses: <2 weeks before Visit 1 OR from Visit 1 till the day of surgery ii) hard contact lenses: <1 month before Visit 1 OR from Visit 1 till the day of surgery iii) therapeutic contact lenses (such as Ortho-K): <3 months before Visit 1 OR from Visit 1 till the day of surgery
2. Corneal disease or pathology, such as corneal scaring or opacity, that precludes transmission of laser wavelength or that distorts laser light
3. Residual, recurrent, or active ocular disease or corneal abnormality (including, but not limited to ocular herpes zoster or simplex, active infections and inflammation)
4. History of ocular herpes simplex or herpes zoster keratitis
5. 3 months before the inclusion have taken systemic medication likely to negatively affect wound healing, such as glucocorticosteroide or antimetabolites
6. Severe dry eye
7. Glaucoma
8. Nystagmus or hemofacial spasm preventing placement of the patient interface
9. Previous corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes
10. Unstable central keratometry readings
11. Mesopic pupil diameter > 8.0 mm
12. Keratometry readings via Sim-K values less than 40.00 D
13. Allergy to medications required in surgery, pre- and post-operative treatment
14. Keratoconus or keratectasia, including patients with suspicion of keratoconus on corneal topography
15. At the time of inclusion, participation in other medical device clinical trials within one month or in drug clinical trials within 3 months
16. Diagnosis of autoimmune disease, connective tissue disease, clinically significant atopic disease, diabetes or AIDS and other acute or chronic illnesses that increases the risk to the subject or confounds the outcomes of this study in the opinion of the study principal investigator
17. Known psychotic disorders associated with delusions (e.g. schizophrenia)
18. Woman who is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
UCDVA (with cycloplegia) | Pre-operative
  The primary outcome is the percentage of eyes that achieve satisfactory Uncorrected Distance Visual Acuity (UCDVA) after CLEAR using the FEMTO LDV Z8, at the time point, when stability of MRSE is reached.
  Satisfactory UCDVA is defined as 20/40, or better, as per Snellen chart lines.
UCDVA (without cycloplegia) | Pre-operative
  The primary outcome is the percentage of eyes that achieve satisfactory Uncorrected Distance Visual Acuity (UCDVA) after CLEAR using the FEMTO LDV Z8, at the time point, when stability of MRSE is reached.
  Satisfactory UCDVA is defined as 20/40, or better, as per Snellen chart lines.
UCDVA | day 1
  The primary outcome is the percentage of eyes that achieve satisfactory Uncorrected Distance Visual Acuity (UCDVA) after CLEAR using the FEMTO LDV Z8, at the time point, when stability of MRSE is reached.
  Satisfactory UCDVA is defined as 20/40, or better, as per Snellen chart lines.
UCDVA | 1 week
  The primary outcome is the percentage of eyes that achieve satisfactory Uncorrected Distance Visual Acuity (UCDVA) after CLEAR using the FEMTO LDV Z8, at the time point, when stability of MRSE is reached.
  Satisfactory UCDVA is defined as 20/40, or better, as per Snellen chart lines.
UCDVA | 1 month
  The primary outcome is the percentage of eyes that achieve satisfactory Uncorrected Distance Visual Acuity (UCDVA) after CLEAR using the FEMTO LDV Z8, at the time point, when stability of MRSE is reached.
  Satisfactory UCDVA is defined as 20/40, or better, as per Snellen chart lines.
UCDVA | 3 months
  The primary outcome is the percentage of eyes that achieve satisfactory Uncorrected Distance Visual Acuity (UCDVA) after CLEAR using the FEMTO LDV Z8, at the time point, when stability of MRSE is reached.
  Satisfactory UCDVA is defined as 20/40, or better, as per Snellen chart lines.
UCDVA | 6 months
  The primary outcome is the percentage of eyes that achieve satisfactory Uncorrected Distance Visual Acuity (UCDVA) after CLEAR using the FEMTO LDV Z8, at the time point, when stability of MRSE is reached.
  Satisfactory UCDVA is defined as 20/40, or better, as per Snellen chart lines.
UCDVA | 9 months
  The primary outcome is the percentage of eyes that achieve satisfactory Uncorrected Distance Visual Acuity (UCDVA) after CLEAR using the FEMTO LDV Z8, at the time point, when stability of MRSE is reached.
  Satisfactory UCDVA is defined as 20/40, or better, as per Snellen chart lines.
UCDVA | 12 months
  The primary outcome is the percentage of eyes that achieve satisfactory Uncorrected Distance Visual Acuity (UCDVA) after CLEAR using the FEMTO LDV Z8, at the time point, when stability of MRSE is reached.
  Satisfactory UCDVA is defined as 20/40, or better, as per Snellen chart lines.

SECONDARY OUTCOMES:
Stability of MRSE | Assessed at 3 months, 6 months, 9 months and 12 months post surgery.
  The percentage of eyes with:
  * a change of less than or equal to 1.00 D of MRSE between two refractions
  * a change of less than or equal to 0.50 D of MRSE between two refractions will be reported for the corresponding time period.
Predictability of MRSE | Up to 12 months
  Percentage of eyes achieving MRSE within ± 1.00 D and within ± 0.50 D of the intended outcome at the point at which MRSE stability is achieved.
Efficacy Index | Up to 12 months
  Efficacy Index is defined as UCDVA at the time point, when stability of MRSE is reached, divided by CDVA at baseline:
  (UCDVA VX /CDVA V1). Note: "X" corresponds to the visit, when stability of MRSE will have been reached.
  The Efficacy Index being above the efficacy cut-off level 0.8 indicates loss of less than two lines of UCDVA
Stability of MRCYL | Assessed at 3 months, 6 months, 9 months and 12 months post surgery.
  The stability of the manifest refractive cylinder (MRCYL) will be evaluated for the whole set of eyes treated for astigmatic myopia. The following statistics for the change in the MRCYL between two consecutive post-operative follow-up visits will be recorded:
  • percentage of eyes with a change in MRCYL within ±1.0 D and ±0.5 D
  Stability analyses will be performed on the eyes that had every follow-up exam from 1- month up to the stability time point (the Consistent Cohort), as well as on the eyes that had 2 consecutive post-op exams, but not necessarily every follow-up exam
Predictability of MRCYL | Up to 12 months
  Percentage of eyes achieving MRCYL within ± 1.00 D of the intended outcome, and within ± 0.50 D of the intended outcome at the point at which stability of MRSE is achieved.
Vector analysis (IRC) | Pre-operative
  Intended Refractive Correction Vector (IRC) IRC = Preoperative cylinder - Target (attempted) cylinder
Vector analysis (SIRC) | Assessed at 3 months, 6 months, 9 months and 12 months post surgery.
  Assessment of change in the Surgically Induced Refractive Correction Vector (SIRC) during follow up; assessed until the MRSE stability is reached.
  SIRC = Preoperative cylinder - Postoperative cylinder
Vector analysis (EV) | Assessed at 3 months, 6 months, 9 months and 12 months post surgery.
  Assessment of change in the Error Vector during follow up; assessed until the MRSE stability is reached.
  Error Vector (EV) EV = IRC - SIRC
Vector analysis (CR) | Assessed at 3 months, 6 months, 9 months and 12 months post surgery.
  Assessment of change in the Correction Rate during follow up; assessed until the MRSE stability is reached.
  Correction Ratio (CR) CR = magnitude of SIRC / magnitude of IRC
Vector analysis (ER) | Assessed at 3 months, 6 months, 9 months and 12 months post surgery.
  Assessment of change in the Error Ratio during follow up; assessed until the MRSE stability is reached.
  Error Ratio (ER) ER = magnitude of EV/ magnitude of IRC
Safety Index | Up to 12 months
  Safety Index defined as CDVA at the time point, when the stability of MRSE is reached, divided by CDVA at baseline (CDVA VX / CDVA V1).
Number of Adverse Events observed in the study | Up to 12 months.
  Complications, including all related (Serious) Adverse Events, during surgery day and follow-up.
Number of Device defects observed in the study | Up to 12 months
  Number of device defects observed during the clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Shi-hao Chen, MD, Principal Investigator — Eye Hospital, WMU
Locations (4):
- China (4):
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Guangzhou Aier Eye Hospital, Guangzhou, Guangdong
  - Ineye Hospital of Chengdu University of TCM, Chengdu, Sichuan
  - Eye Hospital, WMU, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No